CLINICAL TRIAL: NCT07364448
Title: An Open-label, Single-arm Clinical Study to Evaluate the Safety of Hydronidone Capsules in Patients With Liver Fibrosis
Brief Title: A Study to Evaluate the Safety of Hydronidone Capsules in Patients With Liver Fibrosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KDN-F351-202601
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepatitis B With Hepatic Fibrosis
Keywords: Chronic Hepatitis B with Hepatic Fibrosis; Hydronidone
MeSH Terms: interventions — hydronidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydronidone Capsule Group (Experimental): All subjects received hydronidone capsules, administered orally three times daily with three capsules per dose, for a total daily treatment dose of 270 mg. The medication was taken half an hour before meals for a total duration of 28 days.
  Interventions: Drug: Hydronidone capsules

INTERVENTIONS:
Drug: Hydronidone capsules — three times a day, 3 capsules each time,

SUMMARY:
This is an open-label, single-arm study designed to collect safety data on hydronidone capsules in patients with chronic hepatitis B virus infection accompanied by liver fibrosis or fatty liver disease accompanied by liver fibrosis .

Approximately 200 subjects will be enrolled, all of whom will receive hydronidone capsules three times daily, with three capsules per dose, resulting in a total daily treatment dose of 270 mg. The medication will be administered orally half an hour before meals for a total of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of signing the informed consent form (ICF), male or female.
* Patients assessed by the investigator as having chronic hepatitis B with hepatic fibrosis or fatty liver disease with fibrosis (including compensated cirrhosis) based on histology, imaging, or laboratory markers, meeting any of the following criteria:

Histologically confirmed diagnosis of hepatic fibrosis (F2 or above);

Endoscopy showing esophageal or gastric varices or ectopic gastrointestinal varices, excluding non-cirrhotic portal hypertension;

For chronic hepatitis B patients: liver imaging suggestive of fibrotic features, with liver stiffness measurement (LSM) ≥ 8.5 kPa, or Fibrosis-4 Index (FIB-4) ≥ 1.45; Or for non-alcoholic fatty liver disease patients: LSM ≥ 8.5 kPa or FIB-4 ≥ 1.3; Or for alcoholic liver disease patients: LSM ≥ 8.5 kPa.

* Subjects who agree to use effective contraception measures as specified below during their participation in the trial:

Male subjects must consistently employ highly effective contraception methods as described in Appendix 1 from the time of signing the informed consent form until at least 6 months after the last dose of the investigational product.

Female subjects participating in this trial must not be pregnant or lactating and must meet at least one of the following conditions:

1. Be a woman of non-childbearing potential (WONCBP), as defined in Appendix 1;
2. Be a woman of childbearing potential (WOCBP) who consistently uses highly effective contraception methods as described in Appendix 1 from the time of signing the informed consent form until at least 6 months after the last dose of the investigational product, and agrees not to donate eggs for reproductive purposes during this period.

   * The patient voluntarily agrees to participate in this trial, demonstrates good compliance, and has the capacity to understand and sign the informed consent form prior to the study.

Exclusion Criteria:

* At screening, total bilirubin (TBIL) > 3 × upper limit of normal (ULN), or direct bilirubin (DBIL) > 2 × ULN, or alanine aminotransferase (ALT) > 3 × ULN.
* At screening, alpha-fetoprotein (AFP) > 20 μg/L.
* At screening, platelet count (PLT) ≤ 75 × 10⁹/L, or international normalized ratio (INR) > 1.5.
* History of or current clinical diagnosis of decompensated cirrhosis at screening, or imaging showing significant space-occupying lesions in the liver (intrahepatic nodules > 10 mm), or findings suggestive of malignancy.
* Diagnosis of any other malignancy within the past 5 years prior to screening, except for radically resected and non-recurrent skin basal cell carcinoma, cutaneous squamous cell carcinoma, superficial bladder cancer, carcinoma in situ of the cervix (excluding the cervical cancer cohort), localized prostate cancer, or other carcinomas in situ.
* Use of interferon within 3 months prior to screening.
* Concurrent severe diseases of the cardiovascular, pulmonary, renal, endocrine, neurological, digestive, or hematopoietic systems, or psychiatric disorders.
* Planned participation in other interventional clinical trials during the study period.
* Participation in any other clinical trials within 3 months prior to screening.
* Pregnant and/or lactating women.
* Other conditions deemed unsuitable for inclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Any adverse events occurring in study participants following drug administration. | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin University First Hospital, Jilin, Changchun, China